CLINICAL TRIAL: NCT02809534
Title: A Single Group, Open Label, Single-center Clinical Trial to Assess the Efficacy and Safety of Anlotinib in Patients With Hepatocellular Carcinoma (ALTER0802)
Brief Title: A Study of Anlotinib in Patients With Hepatocellular Carcinoma
Acronym: ALTER0802
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTN-08-II
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: Anlotinib; AL3818
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anlotinib (Experimental): Anlotinib QD po and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: Anlotinib

INTERVENTIONS:
Drug: Anlotinib — Anlotinib p.o. qd

SUMMARY:
To assess the primary effects and safety of Anlotinib with placebo in patients with Hepatocellular Carcinoma(HCC).

ELIGIBILITY:
Inclusion Criteria:

* Conform to the clinical diagnosis standard strictly or histological or cytological confirmation of hepatocellular carcinoma who cannot benefit from treatments of ablative therapy
* Liver function status Child-Pugh Class A or B (score≤8)
* Enroll 2 group patients：Group A：No history of systematic chemotherapy/target therapy.Group B:Failed with Sorafenib(Last Sorafenib Therapy≥4 weeks )
* Last Therapy≥4 weeks (such as surgery, PCI,ablation, radiotherapy)，and the wound healing.Patients with adjuvant chemotherapy, last chemotherapy ≥6m
* At least one measurable lesion (by RECIST1.1)
* 18-75 years,ECOG PS:0-1,Life expectancy of more than 3 months
* Main organs function is normal
* Women of childbearing potential should agree to use and utilize an adequate method of contraception (such as intrauterine device，contraceptive and condom) throughout treatment and for at least 6 months after study is stopped；the result of serum or urine pregnancy test should be negative within 7 days prior to study enrollment，and the patients required to be non-lactating；Man participants should agree to use and utilize an adequate method of contraception throughout treatment and for at least 6 months after study is stopped
* Patients should participate in the study voluntarily and sign informed consent

Exclusion Criteria:

* Diagnosed with cholangiocellular carcinoma, mixed cell carcinoma and fibrolamellar hepatocellular carcinoma
* History of other malignancy (except for non-melanoma skin cancer, cervix in situ carcinoma)
* Liver function status Child-Pugh Class C (score>9),with malignant ascites
* HBV-DNA>2000IU/mL
* History of liver transplantation or prepare for it
* Patients with any severe and/or unable to control diseases，including：

  1. Blood pressure unable to be controlled ideally(systolic pressure≥150 mmHg，diastolic pressure≥100 mmHg);
  2. Patients with Grade 1 or higher myocardial ischemia, myocardial infarction or malignant arrhythmias(including QT≥480ms) and patients with Grade 1 or higher congestive heart failure (NYHA Classification);
  3. Patients with active or unable to control serious infections;
  4. Patients with poorly controlled diabetes (fasting blood glucose(FBG)>10mmol/L)
  5. Urine protein ≥ ++，and 24-hour urinary protein excretion>1.0 g confirmed
* Patients with arterial or venous thromboembolic events occurred within 6 months, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis and pulmonary embolism
* Patients with drug abuse history and unable to get rid of or Patients with mental disorders
* Imaging showed tumors have involved important blood vessels or by investigators determine likely during the follow-up study and cause fatal hemorrhage
* Patients participated in other anticancer drug clinical trials within 4 weeks
* History of immunodeficiency
* Patients with concomitant diseases which could seriously endanger their own safety or could affect completion of the study according to investigators' judgment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
12-week Progression-free survival rate(PFR 12w) | From randomization，each 42 days up to PD or death(up to 24 months)

SECONDARY OUTCOMES:
Time to Progression(TTP) | From randomization，each 42 days up to PD or death(up to 24 months)
24-week Progression-free survival rate(PFR 24w) | From randomization，each 42 days up to PD or death(up to 24 months)
Serum Alpha-Fetoprotein level (AFP) | From randomization up to 24 months
Overall Survival (OS) | From randomization until death (up to 24 months)
Objective Response Rate (ORR) | each 42 days up to intolerance the toxicity or PD (up to 24 months)
Disease Control Rate (DCR) | each 42 days up to intolerance the toxicity or PD (up to 24 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided